CLINICAL TRIAL: NCT01569139
Title: Comparison of the Information Recorded in the Myocardial Ischaemia National Audit Project, the General Practice Research Database and Hospital Episode Statistics: a CALIBER Study
Brief Title: Comparison of Information Recorded in MINAP, GPRD and HES: a CALIBER Study
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University College, London (Other); General Practice Research Database (Other Government)
Responsible Party: Principal Investigator, Emily Herrett, Research Degree Student, London School of Hygiene and Tropical Medicine
Other Study IDs: Validation of CALIBER linkage; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome)
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Infarction
Keywords: Validation; Concordance; Myocardial infarction; Myocardial Ischaemia National Audit Project; General Practice Research Database; Hospital Episode Statistics; ONS mortality
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- GPRD MI: Myocardial infarction, as identified in the GPRD data.
- MINAP MI: Myocardial infarction, as identified in MINAP data.
- HES MI: Myocardial infarction, as identified in HES data.

SUMMARY:
Medical information is increasingly processed electronically. This study will describe the similarities and differences in the data recorded by different databases of electronic healthcare database. These will include the General Practice Research Database (GPRD) and the Myocardial Ischaemia National Audit Project (MINAP) and hospital episode statistics (HES).

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

Specific aims are as follows:

1. To validate the linkage between the three databases (General Practice Research Database (GPRD), Myocardial Ischaemia National Audit Project (MINAP), Hospital Episode Statistics (HES)) (checking age, sex and unique identifiers across databases) and establish a cohort of patients with acceptable registration status for further analysis.
2. To describe the ways that MIs are recorded between the three datasets based on the 'best case definition' in each database.

   1. Starting from a 'best case definition' MINAP MI definition (based on the CALIBER phenotype algorithm, which itself is based on the international definition of MI), to examine the way in which the MINAP MI is recorded in GPRD and HES. This analysis will examine STEMI and NSTEMI separately.
   2. Starting from a 'best case definition' algorithm for MI in GPRD (to be decided by GPRD/LSHTM/UCL), to examine the ways in which this MI is recorded in MINAP and HES.
   3. Starting from a 'best case definition' choice of ICD-10 codes for MI in HES, to examine the ways in which this MI is recorded in MINAP and GPRD.
3. To examine predictors of non-concordance between the three datasets.
4. To develop recommendations for a new gold standard definition of MI in each of the databases, based on aims 1-3.

A detailed protocol for this study is available on request. This study has been approved by the Independent Scientific Advisory Committee (ISAC) and by the MINAP Academic Group (MAG).

Study investigators:

R. Boggon, GPRD; Dr S. Denaxas, UCL; Professor H. Hemingway, UCL; E. Herrett, LSHTM; Dr A. Shah, UCL; Professor A. Timmis; Professor T. van Staa, GPRD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Patients in GPRD practices which are deemed "up to standard" by GPRD criteria
* Patients in GPRD whose practice agreed to be linked to the MINAP and HES datasets.
* Patients whose records are deemed "acceptable" by GPRD criteria
* Patients whose age and sex, as recorded in GPRD is the same as that recorded in HES and MINAP.
* Patients with evidence of myocardial infarction in one of the datasets (HES, MINAP, GPRD, ONS) between 1st January 2003 and 6th August 2009.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of "acceptable" patients registered at those GPRD practices that agreed to the linkage with MINAP and HES, whose practices are "up to standard" according to GPRD criteria. Practices taking part in the GPRD are chosen to be representative of UK practices, and 98% of people in the UK are registered with a GP. Therefore the GPRD should be a representative sample of the UK population.
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - London School of Hygiene and Tropical Medicine, London
  - General Practice Research Database, London
  - University College, London, London

REFERENCES:
- [Derived] Herrett E, Shah AD, Boggon R, Denaxas S, Smeeth L, van Staa T, Timmis A, Hemingway H. Completeness and diagnostic validity of recording acute myocardial infarction events in primary care, hospital care, disease registry, and national mortality records: cohort study. BMJ. 2013 May 20;346:f2350. doi: 10.1136/bmj.f2350. PMID 23692896